CLINICAL TRIAL: NCT01473524
Title: A Phase 3, Double-Blind, Placebo-Controlled Trial and Long-Term Safety Extension of Obeticholic Acid in Patients With Primary Biliary Cirrhosis
Brief Title: Phase 3 Study of Obeticholic Acid in Patients With Primary Biliary Cirrhosis
Acronym: POISE
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Intercept Pharmaceuticals (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 747-301
Record Dates: First submitted 2011-11-14; First posted 2011-11-17 (Estimated); Results first posted 2017-02-13 (Actual); Last update posted 2021-05-06 (Actual); Status verified 2021-04

CONDITIONS: Primary Biliary Cirrhosis
Keywords: Primary Biliary Cholangitis; Primary Biliary Cirrhosis; PBC; Cirrhosis; Liver
MeSH Terms: conditions — Liver Cirrhosis, Biliary; Fibrosis | interventions — obeticholic acid

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (4):
- DB OCA 5-10 mg (Experimental): OCA 5 milligram (mg) for 6 months and then titrating up to 10 mg based on tolerability and response for remaining 6 months of the DB phase.
  Interventions: Drug: Obeticholic Acid (OCA)
- DB OCA 10 mg (Experimental): OCA 10 mg for 12 months during the DB phase.
  Interventions: Drug: Obeticholic Acid (OCA)
- DB Placebo (Placebo Comparator): Matching placebo for 12 months during the DB phase.
  Interventions: Drug: Placebo
- LTSE OCA (Experimental): After completion of the 12-month DB phase all participants were offered the opportunity to enter an open-label LTSE for up to 5 years beginning at 5 mg OCA. Initially, participants were allowed to titrate to doses up to 25 mg, however, the maximum dose was then limited to 10 mg. Participants who were previously titrated above 10 mg OCA daily were down-titrated to ≤10 mg OCA daily.
  Interventions: Drug: Obeticholic Acid (OCA)

INTERVENTIONS:
Drug: Obeticholic Acid (OCA) — OCA was administered orally once daily and provided in tablet form in 2 strengths: 5 mg and 10 mg.
  Other Names: 6α-ethyl chenodeoxycholic acid (6-ECDCA); INT-747
  Arms: DB OCA 10 mg; DB OCA 5-10 mg; LTSE OCA
Drug: Placebo — Matching placebo tablets were administered orally once daily.
  Arms: DB Placebo

SUMMARY:
The main objectives of the study were to assess the effects of Obeticholic Acid (OCA) on serum alkaline phosphatase (ALP) and total bilirubin, together as a composite endpoint and on safety in participants with primary biliary cirrhosis (PBC).

DETAILED DESCRIPTION:
The study included 2 phases: a 12-month randomized, double-blind (DB), placebo-controlled, parallel group phase, followed by a long-term safety extension (LTSE) phase up to 5 years. Participants from the 12-month DB phase, including those who received placebo, were eligible to participate in the open-label LTSE phase. The Month 12 visit from the DB phase served as the Day 1 visit of the LTSE phase. After completion of the 12-month DB phase all participants were offered the opportunity to enter an open-label LTSE for up to 5 years beginning at 5 mg OCA.

Data for the LTSE phase is reported by the randomized dose group assigned in the DB phase.

ELIGIBILITY:
Inclusion Criteria:

1. Definite or probable PBC diagnosis (consistent with American Association for the Study of Liver Disease [AASLD] and European Association for Study of the Liver [EASL] Practice Guidelines; [Lindor 2009; EASL 2009]), as demonstrated by the presence of ≥ 2 of the following 3 diagnostic factors:

   * History of elevated alkaline phosphatase (ALP) levels for at least 6 months
   * Positive antimitochondrial antibodies (AMA) titer or if AMA negative or in low titer (<1:80) PBC specific antibodies (anti-GP210 and/or anti-SP100 and/or antibodies against the major M2 components (pyruvate dehydrogenase complex-E2 [PDC-E2], 2-oxo-glutaric acid dehydrogenase complex)
   * Liver biopsy consistent with PBC
2. At least 1 of the following qualifying biochemistry values:

   * ALP ≥ 1.67x upper limit of normal (ULN)
   * Total bilirubin > ULN but < 2x ULN
3. Age ≥ 18 years
4. Taking ursodeoxycholic acid (UDCA) for at least 12 months (stable dose for ≥ 3 months) prior to Day 0, or unable to tolerate UDCA (no UDCA for ≥ 3 months) prior to Day 0.
5. Contraception: Female participants must be postmenopausal, surgically sterile, or if premenopausal, be prepared to use ≥ 1 effective (≤ 1% failure rate) method of contraception during the trial and for 30 days after the end of treatment (EOT) visit. Effective methods of contraception are considered to be:

   * Hormonal (for example, contraceptive pill, patch, intramuscular implant or injection); or
   * Double barrier method, that is, (a) condom (male or female) or (b) diaphragm, with spermicide; or
   * Intrauterine device (IUD); or
   * Vasectomy (partner); or
   * Sexual abstinence
6. Must provide written informed consent and agree to comply with the trial protocol.

Exclusion Criteria:

1. History or presence of other concomitant liver diseases including:

   * Hepatitis C virus (HCV) infection; participants with active hepatitis B (HBV) infection will be excluded, however, participants who have seroconverted (hepatitis B surface antigen [Hbs Ag] and hepatitis B e antigen [Hbe Ag] negative) may be included after consultation with the medical monitor.
   * Primary sclerosing cholangitis (PSC)
   * Alcoholic liver disease
   * Definite autoimmune liver disease or overlap hepatitis
   * Nonalcoholic steatohepatitis (NASH)
   * Gilbert's Syndrome (due to interpretability of bilirubin levels)
2. Presence of clinical complications of PBC or clinically significant hepatic decompensation, including:

   * History of liver transplantation, current placement on a liver transplant list or current Model for End Stage Liver Disease (MELD) score ≥ 15
   * Portal hypertension with complications, including: known gastric or large esophageal varices, poorly controlled or diuretic resistant ascites, history of variceal bleeds or related therapeutic or prophylactic interventions (for example, beta blockers, insertion of variceal bands or transjugular intrahepatic portosystemic shunt [TIPS]), or hepatic encephalopathy
   * Cirrhosis with complications, including history or presence of: spontaneous bacterial peritonitis, hepatocellular carcinoma, bilirubin > 2x ULN
   * Hepatorenal syndrome (type I or II) or Screening serum creatinine > 2 mg/deciliter dL) (178 micromole [µmol])/liter [L])
3. Participants with severe pruritus or those requiring systemic treatment for pruritus (for example, with bile acid sequestrants [BAS] or rifampicin) within 2 months of Day 0 will be excluded
4. Administration of the following medications is prohibited as specified below:

   * Prohibited 6 months prior to Day 0 and throughout the trial (that is, to last dose and/or EOT): azathioprine, colchicine, cyclosporine, methotrexate, mycophenolate mofetil, pentoxifylline; fenofibrate or other fibrates; budesonide and other systemic corticosteroids; potentially hepatotoxic drugs (including α-methyl-dopa, sodium valproic acid, isoniazide, or nitrofurantoin)
   * Prohibited 12 months prior to Day 0 and throughout the trial (that is, to last dose and/or EOT): antibodies or immunotherapy directed against interleukins or other cytokines or chemokines
5. Participants who have previously participated in a clinical trial of OCA will not be allowed to participate
6. History or presence of clinically concerning cardiac arrhythmias likely to affect survival during the trial, or prolongation of Screening (pretreatment) QT or QTc interval of > 500 milliseconds (msec)
7. If female: known pregnancy, or has a positive urine pregnancy test (confirmed by a positive serum pregnancy test), or lactating
8. Known history of human immunodeficiency virus (HIV) infection
9. Presence of any other disease or condition that is interfering with the absorption, distribution, metabolism, or excretion of drugs including bile salt metabolism in the intestine. Participants with inflammatory bowel disease or who have undergone gastric bypass procedures will be excluded (gastric lap band is acceptable).
10. Medical conditions that may cause nonhepatic increases in ALP (for example, Paget's disease) or which may diminish life expectancy to < 2 years, including known cancers (except carcinomas in situ or other stable, relatively benign conditions such as chronic lymphatic leukemia)
11. Other clinically significant medical conditions that are not well controlled or for which medication needs are anticipated to change during the trial
12. Anticipated changes to current concomitant medications during the course of the trial
13. History of alcohol abuse, defined as consumption of more than 210 mL of alcohol per week (that is, the equivalent of fourteen 4-ounce (125 mL) glasses of wine or fourteen 12 ounce cans/bottles of beer), or other substance abuse within 1 year prior to Day 0
14. Participation in another investigational drug, biologic, or medical device trial within 30 days prior to Screening
15. History of noncompliance with medical regimens, or participants who are considered to be potentially unreliable
16. Blood or plasma donation within 30 days prior to Day 0
17. Mental instability or incompetence, such that the validity of informed consent or compliance with the trial is uncertain

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 217 (Actual)
Dates: Start 2012-01; Primary Completion 2013-12 (Actual); Study Completion 2018-12-17 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Christian Weyer, MD, Study Chair — Intercept Pharmaceuticals, Inc.
Locations (59):
- United States (15):
  - UC Davis Medical Center, Sacramento, California
  - Scripps Clinic, San Diego, California
  - University of Colorado, Denver, Aurora, Colorado
  - University of Chicago, Chicago, Illinois
  - Indiana University School of Medicine, Indianapolis, Indiana
  - Henry Ford Health System, Detroit, Michigan
  - St. Louis University, St Louis, Missouri
  - Beth Israel Medical Center, New York, New York
  - Duke University Medical Center, Durham, North Carolina
  - University of Texas Southwestern Medical Center, Dallas, Texas
  - Baylor College of Medicine, Houston, Texas
  - Liver Institute of Virginia, Newport News, Virginia
  - Liver Institute of Virginia, Richmond, Virginia
  - Virginia Commonwealth University/McGuire DVAMC, Richmond, Virginia
  - Swedish Medical Center, Seattle, Washington
- Australia (3):
  - Royal Prince Alfred Hospital, Camperdown, New South Wales
  - Austin Hospital, Heidelberg, Victoria
  - The Alfred Hospital, Melbourne, Victoria
- Austria (2):
  - Medizinische Universität Innsbruck, Innsbruck
  - Medizinische Universität Wien, Vienna
- UZ Leuven, Leuven, Belgium
- Canada (2):
  - Toronto Western Hospital Liver Centre, Toronto, Ontario
  - CHUM Hôpital St-Luc, Montreal, Quebec
- Hopital Haut-Leveque, Pessac, France
- Germany (10):
  - Universitätsklinikum Aachen, Aachen
  - Friedrich-Alexander-Universität Erlangen, Erlangen
  - Klinikum der Johann-Wolfgang Goethe Universität Frankfurt am Main, Frankfurt am Main
  - Universitätsklinikum Hamburg Eppendorf, Hamburg
  - Medizinische Hochschule Hannover, Hanover
  - Medizinische Universitätsklinik, Heidelberg
  - Gastroenterologische Gemeinschaftspraxis, Dres. Felten / Hartmann / Hüppe, Herne
  - Universitätsklinikum des Saarlandes, Homburg
  - Universitätsklinikum Leipzig, Leipzig
  - LMU Klinikum der Universität München, München
- Italy (4):
  - Dip. Medicina Clinica - Università di Bologna, Bologna
  - Dip. Medicina Clinica- Università di Bologna, Bologna
  - Azienda Ospedaliera di Padova - Gastroenterologia, Padua
  - Istituto Clinico Humanitas, Rozzano (MI)
- Netherlands (4):
  - VUmc Amsterdam, Amsterdam
  - AMC Amsterdam, Amsterdam
  - UMC St. Radboud, Nijmegen, Nijmegen
  - UMC Utrecht, Utrecht
- Poland (5):
  - All-Medicus, Katowice
  - Klinika Gastroenterologii i Hepatologii SP CSK im. prof. K. Gibinskiego SUM, Katowice
  - Samodzielny Publiczny Szpital Kliniczny nr 4 w Lublinie, Lublin
  - Niepubliczny Zakład Opieki Zdrowotnej "SONOMED", Szczecin
  - Centrum Onkologii - Instytut im. Marii Skłodowskiej - Curie, Klinika Gastroenterologii, Warsaw
- Spain (2):
  - Hospital Vall d'Hebron, Barcelona
  - Hospital Clinic de Barcelona, Barcelona
- Sahlgrenska University Hospital, Gothenburg, Sweden
- United Kingdom (9):
  - Queen Elizabeth Hospital, Birmingham
  - Bristol Royal Infirmary, Bristol
  - Ninewells Hospital Dundee, Dundee
  - Forth Valley Royal Hospital, Larbert
  - The Royal Free Hospital, London
  - Manchester Royal Infirmary, Manchester
  - Institute of Cellular Medicine, Newcastle University, Newcastle upon Tyne
  - Nottingham University Hospitals NHS Trust, Nottingham
  - Oxford University Hospitals Trust, Oxford

REFERENCES:
- [Background] Lindor KD, Gershwin ME, Poupon R, Kaplan M, Bergasa NV, Heathcote EJ; American Association for Study of Liver Diseases. Primary biliary cirrhosis. Hepatology. 2009 Jul;50(1):291-308. doi: 10.1002/hep.22906. No abstract available. PMID 19554543
- [Result] Nevens F, Andreone P, Mazzella G, Strasser SI, Bowlus C, Invernizzi P, Drenth JP, Pockros PJ, Regula J, Beuers U, Trauner M, Jones DE, Floreani A, Hohenester S, Luketic V, Shiffman M, van Erpecum KJ, Vargas V, Vincent C, Hirschfield GM, Shah H, Hansen B, Lindor KD, Marschall HU, Kowdley KV, Hooshmand-Rad R, Marmon T, Sheeron S, Pencek R, MacConell L, Pruzanski M, Shapiro D; POISE Study Group. A Placebo-Controlled Trial of Obeticholic Acid in Primary Biliary Cholangitis. N Engl J Med. 2016 Aug 18;375(7):631-43. doi: 10.1056/NEJMoa1509840. PMID 27532829
- [Result] Trauner M, Nevens F, Shiffman ML, Drenth JPH, Bowlus CL, Vargas V, Andreone P, Hirschfield GM, Pencek R, Malecha ES, MacConell L, Shapiro D. Long-term efficacy and safety of obeticholic acid for patients with primary biliary cholangitis: 3-year results of an international open-label extension study. Lancet Gastroenterol Hepatol. 2019 Jun;4(6):445-453. doi: 10.1016/S2468-1253(19)30094-9. Epub 2019 Mar 26. PMID 30922873
- [Derived] Harms MH, Hirschfield GM, Floreani A, Mayo MJ, Pares A, Liberman A, Malecha ES, Pencek R, MacConell L, Hansen BE. Obeticholic acid is associated with improvements in AST-to-platelet ratio index and GLOBE score in patients with primary biliary cholangitis. JHEP Rep. 2020 Sep 29;3(1):100191. doi: 10.1016/j.jhepr.2020.100191. eCollection 2021 Feb. PMID 33319187
- [Derived] Bowlus CL, Pockros PJ, Kremer AE, Pares A, Forman LM, Drenth JPH, Ryder SD, Terracciano L, Jin Y, Liberman A, Pencek R, Iloeje U, MacConell L, Bedossa P. Long-Term Obeticholic Acid Therapy Improves Histological Endpoints in Patients With Primary Biliary Cholangitis. Clin Gastroenterol Hepatol. 2020 May;18(5):1170-1178.e6. doi: 10.1016/j.cgh.2019.09.050. Epub 2019 Oct 10. PMID 31606455
- [Derived] Mousa HS, Lleo A, Invernizzi P, Bowlus CL, Gershwin ME. Advances in pharmacotherapy for primary biliary cirrhosis. Expert Opin Pharmacother. 2015 Apr;16(5):633-43. doi: 10.1517/14656566.2015.998650. Epub 2014 Dec 29. PMID 25543678

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Recruitment into hospitals and physicians' clinics started January 2012 and completed December 2012.
Pre-assignment Details: Screening interim allowed for pre-randomization eligibility assessment of 1 to 8 weeks.
  A total of 217 participants were randomized into the double-blind phase of the study, however, 216 received treatment with study drug. One randomized participant discontinued prior to receiving any study drug.
Groups:
- DB OCA 5-10 mg: Obeticholic acid (OCA) 5 mg for 6 months and then titrating up to 10 mg based on tolerability and response for remaining 6 months of the double-blind (DB) phase.
- DB OCA 10 mg: OCA 10 mg for 12 months during DB phase.
- DB Placebo: Matching placebo for 12 months in the DB phase.
- LTSE OCA (DB OCA 5-10 mg): Participants previously receiving OCA 5 to 10 mg in the DB phase received OCA in the open-label long-term safety extension (LTSE) phase for up to 5 years beginning at 5 mg, and then the dose could be titrated up. Initially, participants were allowed to titrate to doses up to 25 mg, however, the maximum dose was then limited to 10 mg.
- LTSE OCA (DB OCA 10 mg): Participants previously receiving OCA 10 mg in the DB phase received OCA in the open-label LTSE phase for up to 5 years beginning at 5 mg, and then the dose could be titrated up. Initially, participants were allowed to titrate to doses up to 25 mg, however, the maximum dose was then limited to 10 mg.
- LTSE OCA (DB Placebo): Participants previously receiving placebo in the DB phase received OCA in the open-label LTSE phase for up to 5 years beginning at 5 mg, and then the dose could be titrated up. Initially, participants were allowed to titrate to doses up to 25 mg, however, the maximum dose was then limited to 10 mg.
Period: DB Phase
Arm/Group | DB OCA 5-10 mg | DB OCA 10 mg | DB Placebo | LTSE OCA (DB OCA 5-10 mg) | LTSE OCA (DB OCA 10 mg) | LTSE OCA (DB Placebo)
Started | 71 | 73 | 73 | 0 | 0 | 0
Received at Least 1 Dose of Study Drug | 70 | 73 | 73 | 0 | 0 | 0
Completed | 64 | 64 | 70 | 0 | 0 | 0
Not Completed | 7 | 9 | 3 | 0 | 0 | 0
Not completed — Adverse Event | 4 | 8 | 2 | 0 | 0 | 0
Not completed — Death | 1 | 0 | 0 | 0 | 0 | 0
Not completed — Withdrawal by Subject | 2 | 1 | 1 | 0 | 0 | 0
Period: LTSE Phase
Arm/Group | DB OCA 5-10 mg | DB OCA 10 mg | DB Placebo | LTSE OCA (DB OCA 5-10 mg) | LTSE OCA (DB OCA 10 mg) | LTSE OCA (DB Placebo)
Started | 0 | 0 | 0 | 63 (One participant in the double-blind OCA 5-10 mg group did not enroll in the LTSE phase.) | 64 | 66 (Four participants in the double-blind placebo group did not enroll in the LTSE phase.)
Received at Least 1 Dose of OCA in LTSE | 0 | 0 | 0 | 63 | 64 | 66
Completed | 0 | 0 | 0 | 54 | 47 | 45
Not Completed | 0 | 0 | 0 | 9 | 17 | 21
Not completed — Withdrawal by Subject | 0 | 0 | 0 | 3 | 3 | 6
Not completed — Death | 0 | 0 | 0 | 0 | 1 | 0
Not completed — Adverse Event of Pruritus | 0 | 0 | 0 | 1 | 5 | 2
Not completed — Other Clinical/ Laboratory Adverse Event | 0 | 0 | 0 | 2 | 4 | 6
Not completed — Lost to Follow-up | 0 | 0 | 0 | 1 | 3 | 2
Not completed — Principal Investigator Decision | 0 | 0 | 0 | 1 | 1 | 3
Not completed — Liver Transplantation | 0 | 0 | 0 | 0 | 0 | 1
Not completed — Pregnancy | 0 | 0 | 0 | 1 | 0 | 0
Not completed — Protocol Violation | 0 | 0 | 0 | 0 | 0 | 1

BASELINE CHARACTERISTICS:
Population: Intent-to-treat Population: All participants who were randomized and received at least 1 dose of study drug.
Groups:
- DB OCA 5-10 mg: OCA 5 mg for 6 months and then titrating up to 10 mg based on tolerability and response for remaining 6 months of the DB phase.
  After completion of the 12-month DB phase participants were offered the opportunity to enter an open-label LTSE for up to 5 years beginning at 5 mg OCA, and then the dose could be titrated up. Initially, participants were allowed to titrate to doses up to 25 mg, however, the maximum dose was then limited to 10 mg.
- DB OCA 10 mg: OCA 10 mg 12 months during the DB phase. After completion of the 12-month DB phase participants were offered the opportunity to enter an open-label LTSE for up to 5 years beginning at 5 mg OCA, and then the dose could be titrated up. Initially, participants were allowed to titrate to doses up to 25 mg, however, the maximum dose was then limited to 10 mg.
- DB Placebo: Matching placebo for 12 months during the DB phase. After completion of the 12-month DB phase participants were offered the opportunity to enter an open-label LTSE for up to 5 years beginning at 5 mg OCA, and then the dose could be titrated up. Initially, participants were allowed to titrate to doses up to 25 mg, however, the maximum dose was then limited to 10 mg.
- Total: Total of all reporting groups
Arm/Group | DB OCA 5-10 mg | DB OCA 10 mg | DB Placebo | Total
Number analyzed (Participants) | 70 | 73 | 73 | 216
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0 | 0
  Between 18 and 65 years | 60 | 56 | 60 | 176
  >=65 years | 10 | 17 | 13 | 40
Age, Continuous [Mean (Standard Deviation); unit: years] | 55.8 (10.53) | 56.2 (11.00) | 55.5 (10.03) | 55.8 (10.48)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 65 | 63 | 68 | 196
  Male | 5 | 10 | 5 | 20
Race/Ethnicity, Customized [Number; unit: participants]
  Asian | 1 | 1 | 1 | 3
  Black or African American | 1 | 1 | 1 | 3
  Other | 1 | 1 | 5 | 7
  White | 67 | 70 | 66 | 203
Region of Enrollment [Number; unit: participants]
  United States | 18 | 19 | 17 | 54
  United Kingdom | 8 | 5 | 9 | 22
  Spain | 4 | 2 | 3 | 9
  Canada | 2 | 2 | 4 | 8
  Austria | 2 | 0 | 1 | 3
  Netherlands | 3 | 7 | 6 | 16
  Sweden | 3 | 1 | 0 | 4
  Belgium | 2 | 9 | 5 | 16
  Poland | 4 | 6 | 4 | 14
  Italy | 11 | 10 | 11 | 32
  Australia | 5 | 1 | 3 | 9
  France | 0 | 0 | 1 | 1
  Germany | 8 | 11 | 9 | 28
Alkaline Phosphatase (U/L) [Mean (Standard Deviation); unit: U/L] | 325.87 (116.238) | 316.34 (103.881) | 327.49 (115.014) | 323.19 (111.375)
Total Bilirubin (umol/L) [Mean (Standard Deviation); unit: umol/L] | 10.192 (5.549) | 11.278 (6.634) | 11.757 (7.227) | 11.088 (6.522)
Direct Bilirubin (umol/L) [Mean (Standard Deviation); unit: umol/L] | 4.398 (4.528) | 4.868 (4.473) | 5.469 (6.214) | 4.919 (5.138)
Alanine Aminotransferase (ALT) (U/L) [Mean (Standard Deviation); unit: U/L] | 61.56 (39.037) | 56.31 (39.741) | 55.99 (30.312) | 57.9 (36.498)
Aspartate Aminotransferase (AST) (U/L) [Mean (Standard Deviation); unit: U/L] | 52.25 (25.289) | 50.49 (31.100) | 48.79 (22.449) | 50.49 (26.456)
Gamma-Glutamyltransferase (GGT) (U/L) [Mean (Standard Deviation); unit: U/L] | 252.83 (167.038) | 261.07 (207.396) | 309.58 (449.356) | 274.79 (302.673)

OUTCOME MEASURES:

1. Primary Outcome: DB Phase: Composite Endpoint Alkaline Phosphatase (ALP) And Total Bilirubin, 10 mg OCA Versus Placebo
Description: Percentage of participants at Month 12 with ALP < 1.67 x upper limit of normal (ULN) and total bilirubin ≤ ULN and ALP decrease of ≥ 15% from baseline.
Time Frame: DB Month 12
Population: Intent-to-Treat Population: All participants who were randomized and received at least 1 dose of study drug.
Measure: Number; unit: percentage of participants
Arm/Group | DB OCA 10 mg | DB Placebo
Number analyzed (Participants) | 73 | 73
percentage of participants | 47 | 10
Statistical Analysis 1: Comparison: DB OCA 10 mg vs DB Placebo; H0: The response rates are equal between placebo and 10 mg OCA. H1: The response rates are different between placebo and 10 mg OCA; Test type: Superiority or Other; p < 0.0001, Cochran-Mantel-Haenszel; Cochran-Mantel-Haenszel (CMH) General Association test stratified by randomization strata factor

2. Primary Outcome: LTSE Phase: Composite Endpoint ALP And Total Bilirubin
Description: Percentage of participants at Months 24, 36, 48, and 60 with ALP < 1.67x ULN and total bilirubin ≤ ULN and ALP decrease of ≥ 15% from baseline. DB Month 12 is the baseline for the LTSE phase.
Time Frame: Baseline (DB Month 12), LTSE Months 24, 36, 48, and 60
Population: All participants who received at least 1 dose of OCA in the open-label safety extension phase and had an assessment at the specified timepoint.
Measure: Number; unit: percentage of participants
Groups:
- LTSE OCA (DB OCA 5-10 mg): Participants previously receiving OCA 5-10 mg in the DB phase received OCA in the open-label LTSE phase for up to 5 years beginning at 5 mg, and then the dose could be titrated up. Initially, participants were allowed to titrate to doses up to 25 mg, however, the maximum dose was then limited to 10 mg.
- Overall LTSE OCA: After completion of the 12-month DB phase all participants were offered the opportunity to enter an open-label LTSE for up to 5 years beginning at 5 mg OCA, and then the dose could be titrated up. Initially, participants were allowed to titrate to doses up to 25 mg, however, the maximum dose was then limited to 10 mg.
Arm/Group | LTSE OCA (DB OCA 5-10 mg) | LTSE OCA (DB OCA 10 mg) | LTSE OCA (DB Placebo) | Overall LTSE OCA
Number analyzed (Participants) | 63 | 64 | 66 | 193
percentage of participants
  Baseline (Double-blind Month 12): number analyzed (Participants) | 63 | 63 | 66 | 192
  Baseline (Double-blind Month 12) | 51 | 56 | 9 | 38
  LTSE Month 12: number analyzed (Participants) | 60 | 59 | 59 | 178
  LTSE Month 12 | 55 | 58 | 41 | 51
  LTSE Month 24: number analyzed (Participants) | 57 | 57 | 52 | 166
  LTSE Month 24 | 60 | 61 | 54 | 58
  LTSE Month 36: number analyzed (Participants) | 56 | 55 | 49 | 160
  LTSE Month 36 | 48 | 51 | 49 | 49
  LTSE Month 48: number analyzed (Participants) | 50 | 53 | 48 | 151
  LTSE Month 48 | 52 | 55 | 60 | 56
  LTSE Month 60: number analyzed (Participants) | 31 | 21 | 24 | 76
  LTSE Month 60 | 48 | 52 | 50 | 50

3. Secondary Outcome: DB Phase: Composite Endpoint ALP And Total Bilirubin, 10 mg Versus Placebo
Description: Percentage of participants at Month 6 with ALP < 1.67x ULN and total bilirubin ≤ ULN and ALP decrease of ≥ 15% from baseline.
Time Frame: DB Month 6
Population: Intent-to-Treat Population: All participants who were randomized and received at least 1 dose of study drug.
Measure: Number; unit: percentage of participants
Groups:
- Double-blind OCA 10 mg: OCA 10 mg for 12 months during the DB phase.
- Double-blind Placebo: Matching placebo for 12 months during the DB phase.
Arm/Group | Double-blind OCA 10 mg | Double-blind Placebo
Number analyzed (Participants) | 73 | 73
percentage of participants | 51 | 7
Statistical Analysis 1: Comparison: Double-blind OCA 10 mg vs Double-blind Placebo; [analysis description as in outcome 1, analysis 1]; Test type: Superiority or Other; p < 0.0001, Cochran-Mantel-Haenszel; Cochran-Mantel-Haenszel (CMH) General Association test stratified by randomization strata factor

4. Secondary Outcome: DB Phase: Composite Endpoint ALP And Total Bilirubin, 5-10 mg Versus Placebo
Description: Percentage of participants at Month 12 with ALP < 1.67x ULN and total bilirubin ≤ ULN and ALP decrease of ≥ 15% from baseline.
Time Frame: DB Month 12
Population: Intent-to-Treat Population: All participants who were randomized and received at least 1 dose of study drug.
Measure: Number; unit: percentage of participants
Groups:
- DB OCA 5-10 mg: OCA 5 mg for 6 months and then titrating up to 10 mg based on tolerability and response for remaining 6 months of the DB phase.
Arm/Group | DB OCA 5-10 mg | DB Placebo
Number analyzed (Participants) | 70 | 73
percentage of participants | 46 | 10
Statistical Analysis 1: Comparison: DB OCA 5-10 mg vs DB Placebo; H0: The response rates are equal between placebo and 5-10 mg OCA. H1: The response rates are different between placebo and 5-10 mg OCA; Test type: Superiority or Other; p < 0.0001, Cochran-Mantel-Haenszel; Cochran-Mantel-Haenszel (CMH) General Association test stratified by randomization strata factor

5. Secondary Outcome: DB Phase: Composite Endpoint ALP And Total Bilirubin, 5-10 mg Versus Placebo
Description: as for outcome 3
Time Frame: DB Month 6
Population: Intent-to-Treat Population: All participants who were randomized and received at least 1 dose of study drug.
Measure: Number; unit: percentage of participants
Arm/Group | DB OCA 5-10 mg | DB Placebo
Number analyzed (Participants) | 70 | 73
percentage of participants | 34 | 7
Statistical Analysis 1: Comparison: DB OCA 5-10 mg vs DB Placebo; [analysis description as in outcome 4, analysis 1]; Test type: Superiority or Other; p < 0.0001, Cochran-Mantel-Haenszel; Cochran-Mantel-Haenszel (CMH) General Association test stratified by randomization strata factor

6. Secondary Outcome: DB Phase: ALP Absolute Change From Baseline To Month 12
Description: Blood samples were evaluated for ALP levels. ALP Absolute Change From Baseline (ALP at Month 12 - ALP at Baseline) is presented.
Time Frame: Baseline, DB Month 12
Population: Intent-to-Treat Population: All participants who were randomized and received at least 1 dose of study drug and had an assessment at the specified timepoint.
Measure: Least Squares Mean (Standard Error); unit: U/L
Groups:
- DB Placebo: Matching placebo during the DB phase.
Arm/Group | DB OCA 5-10 mg | DB OCA 10 mg | DB Placebo
Number analyzed (Participants) | 64 | 62 | 70
U/L | -112.51 (14.36) | -129.90 (14.60) | -14.42 (14.74)
Statistical Analysis 1: Comparison: DB OCA 5-10 mg vs DB Placebo; Test type: Superiority or Other; p < 0.0001, ANCOVA; ANCOVA model with baseline value as a covariate and fixed effects for treatment and randomization strata factor
Statistical Analysis 2: Comparison: DB OCA 10 mg vs DB Placebo; Test type: Superiority or Other; p < 0.0001, ANCOVA; ANCOVA model with baseline value as a covariate and fixed effects for treatment and randomization strata factor

7. Secondary Outcome: DB Phase: Total Bilirubin Absolute Change From Baseline To Month 12
Description: Blood samples were evaluated for bilirubin levels. Total bilirubin absolute change from baseline (total bilirubin at Month 12 - total bilirubin at Baseline) is presented.
Time Frame: Baseline, DB Month 12
Population: as for outcome 6
Measure: Least Squares Mean (Standard Error); unit: umol/L
Arm/Group | DB OCA 5-10 mg | DB OCA 10 mg | DB Placebo
Number analyzed (Participants) | 64 | 62 | 70
umol/L | -0.33 (0.68) | -0.90 (0.71) | 1.98 (0.70)
Statistical Analysis 1: Comparison: DB OCA 5-10 mg vs DB Placebo; Test type: Superiority or Other; p = 0.0004, ANCOVA; ANCOVA model with baseline value as a covariate and fixed effects for treatment and randomization strata factor
Statistical Analysis 2: Comparison: DB OCA 10 mg vs DB Placebo; Test type: Superiority or Other; p < 0.0001, ANCOVA; ANCOVA model with baseline value as a covariate and fixed effects for treatment and randomization strata factor

8. Secondary Outcome: DB Phase: Direct Bilirubin Absolute Change From Baseline To Month 12
Description: Blood samples were evaluated for bilirubin levels. Direct bilirubin absolute change from baseline (direct bilirubin at Month 12 - direct bilirubin at Baseline) is presented.
Time Frame: Baseline, DB Month 12
Population: as for outcome 6
Measure: Least Squares Mean (Standard Error); unit: umol/L
Arm/Group | DB OCA 5-10 mg | DB OCA 10 mg | DB Placebo
Number analyzed (Participants) | 64 | 62 | 70
umol/L | -0.13 (0.52) | -0.49 (0.54) | 1.89 (0.53)
Statistical Analysis 1: Comparison: DB OCA 5-10 mg vs DB Placebo; Test type: Superiority or Other; p < 0.0001, ANCOVA; ANCOVA model with baseline value as a covariate and fixed effects for treatment and randomization strata factor
Statistical Analysis 2: Comparison: DB OCA 10 mg vs DB Placebo; Test type: Superiority or Other; p < 0.0001, ANCOVA; ANCOVA model with baseline value as a covariate and fixed effects for treatment and randomization strata factor

9. Secondary Outcome: DB Phase: Alanine Aminotransferase (ALT) Absolute Change From Baseline To Month 12
Description: Blood samples were evaluated for ALT levels. ALT absolute change from baseline (ALT at Month 12 - ALT at Baseline) is presented.
Time Frame: Baseline, DB Month 12
Population: as for outcome 6
Measure: Least Squares Mean (Standard Error); unit: U/L
Arm/Group | DB OCA 5-10 mg | DB OCA 10 mg | DB Placebo
Number analyzed (Participants) | 64 | 62 | 70
U/L | -21.26 (3.27) | -25.31 (3.35) | -4.95 (3.32)
Statistical Analysis 1: Comparison: DB OCA 5-10 mg vs DB Placebo; Test type: Superiority or Other; p < 0.0001, ANCOVA; ANCOVA model with baseline value as a covariate and fixed effects for treatment and randomization strata factor
Statistical Analysis 2: Comparison: DB OCA 10 mg vs DB Placebo; Test type: Superiority or Other; p < 0.0001, ANCOVA; ANCOVA model with baseline value as a covariate and fixed effects for treatment and randomization strata factor

10. Secondary Outcome: DB Phase: Aspartate Aminotransferase (AST) Absolute Change From Baseline To Month 12
Description: Blood samples were evaluated for AST levels. AST absolute change from baseline (AST at Month 12 - AST at Baseline) is presented.
Time Frame: Baseline, DB Month 12
Population: as for outcome 6
Measure: Least Squares Mean (Standard Error); unit: U/L
Groups:
- DB OCA 5-10 mg: OCA 5 mg for 6 months and then titrating up to 10 mg based on tolerability and response for remaining 12 months of the DB phase.
Arm/Group | DB OCA 5-10 mg | DB OCA 10 mg | DB Placebo
Number analyzed (Participants) | 64 | 62 | 70
U/L | -13.03 (4.17) | -15.00 (4.28) | 1.04 (4.22)
Statistical Analysis 1: Comparison: DB OCA 5-10 mg vs DB Placebo; Test type: Superiority or Other; p = 0.0003, ANCOVA; ANCOVA model with baseline value as a covariate and fixed effects for treatment and randomization strata factor
Statistical Analysis 2: Comparison: DB OCA 10 mg vs DB Placebo; Test type: Superiority or Other; p < 0.0001, ANCOVA; ANCOVA model with baseline value as a covariate and fixed effects for treatment and randomization strata factor

11. Secondary Outcome: DB Phase: Gamma-glutamyltransferase (GGT) Absolute Change From Baseline To Month 12
Description: Blood samples were evaluated for GGT levels. GGT absolute change from baseline (GGT at Month 12 - GGT at Baseline) is presented.
Time Frame: Baseline, DB Month 12
Population: as for outcome 6
Measure: Least Squares Mean (Standard Error); unit: U/L
Arm/Group | DB OCA 5-10 mg | DB OCA 10 mg | DB Placebo
Number analyzed (Participants) | 64 | 62 | 70
U/L | -140.83 (24.70) | -176.66 (25.58) | 6.70 (25.56)
Statistical Analysis 1: Comparison: DB OCA 5-10 mg vs DB Placebo; Test type: Superiority or Other; p < 0.0001, ANCOVA; ANCOVA model with baseline value as a covariate and fixed effects for treatment and randomization strata factor
Statistical Analysis 2: Comparison: DB OCA 10 mg vs DB Placebo; Test type: Superiority or Other; p < 0.0001, ANCOVA; ANCOVA model with baseline value as a covariate and fixed effects for treatment and randomization strata factor

12. Secondary Outcome: LTSE Phase: ALP Levels
Description: Blood samples were evaluated for ALP levels.
Time Frame: LTSE Day 0 and LTSE Months 12, 24, 36, 48, and 60
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: U/L
Arm/Group | LTSE OCA (DB OCA 5-10 mg) | LTSE OCA (DB OCA 10 mg) | LTSE OCA (DB Placebo) | Overall LTSE OCA
Number analyzed (Participants) | 63 | 64 | 66 | 193
U/L
  LTSE Day 0: number analyzed (Participants) | 63 | 63 | 66 | 192
  LTSE Day 0 | 218.69 (100.328) | 191.24 (61.381) | 317.79 (139.666) | 243.75 (118.910)
  LTSE Month 12: number analyzed (Participants) | 60 | 59 | 59 | 178
  LTSE Month 12 | 209.49 (93.157) | 198.68 (75.799) | 226.28 (105.404) | 211.47 (92.439)
  LTSE Month 24: number analyzed (Participants) | 57 | 57 | 52 | 166
  LTSE Month 24 | 195.14 (80.361) | 194.57 (66.593) | 215.99 (83.469) | 201.47 (77.117)
  LTSE Month 36: number analyzed (Participants) | 56 | 55 | 49 | 160
  LTSE Month 36 | 204.52 (68.019) | 214.66 (158.831) | 205.37 (65.206) | 208.27 (107.114)
  LTSE Month 48: number analyzed (Participants) | 50 | 53 | 48 | 151
  LTSE Month 48 | 189.75 (55.929) | 192.00 (59.761) | 198.70 (65.551) | 193.38 (60.170)
  LTSE Month 60: number analyzed (Participants) | 31 | 21 | 24 | 76
  LTSE Month 60 | 200.90 (97.475) | 191.37 (62.404) | 209.38 (82.240) | 200.94 (83.436)

13. Secondary Outcome: LTSE Phase: ALP Change From DB Baseline
Description: Blood samples were evaluated for ALP levels. ALP Change From Baseline (ALP at LTSE Months 12, 24, 36, 48, and 60 - ALP at Baseline) is presented. DB baseline is the mean of all available evaluations prior to DB treatment.
Time Frame: DB Baseline, LTSE Months 12, 24, 36, 48, and 60
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: U/L
Arm/Group | LTSE OCA (DB OCA 5-10 mg) | LTSE OCA (DB OCA 10 mg) | LTSE OCA (DB Placebo) | Overall LTSE OCA
Number analyzed (Participants) | 63 | 64 | 66 | 193
U/L
  Month 12: number analyzed (Participants) | 60 | 59 | 59 | 178
  Month 12 | -106.63 (98.448) | -104.39 (82.496) | -104.36 (83.074) | -105.13 (87.882)
  Month 24: number analyzed (Participants) | 57 | 57 | 52 | 166
  Month 24 | -120.86 (96.614) | -102.52 (79.413) | -100.99 (87.181) | -108.34 (87.980)
  Month 36: number analyzed (Participants) | 56 | 55 | 49 | 160
  Month 36 | -100.98 (109.952) | -84.65 (137.293) | -112.73 (89.661) | -98.96 (114.635)
  Month 48: number analyzed (Participants) | 50 | 53 | 48 | 151
  Month 48 | -118.23 (101.527) | -101.50 (91.335) | -115.51 (106.774) | -111.49 (99.433)
  Month 60: number analyzed (Participants) | 31 | 21 | 24 | 60
  Month 60 | -118.99 (147.126) | -117.49 (95.587) | -119.52 (108.949) | -118.74 (121.391)

ADVERSE EVENTS:
Time Frame: DB Phase: Baseline up to 12 months (1 year). LTSE phase: Baseline (DB Month 12) up to 60 months (5 years).
Groups:
- DB 5-10 mg: OCA 5 mg for 6 months and then titrating up to 10 mg based on tolerability and response for remaining 6 months of the DB phase.
- LTSE OCA (DB OCA 5-10 mg): Participants previously receiving OCA 5 to 10 mg in the DB phase received OCA in the open-label LTSE phase for up to 5 years beginning at 5 mg, and then the dose could be titrated up. Initially, participants were allowed to titrate to doses up to 25 mg, however, the maximum dose was then limited to 10 mg.
- LTSE OCA (DB 10 mg): Participants previously receiving OCA 10 mg in the DB phase received OCA in the open-label LTSE phase for up to 5 years beginning at 5 mg, and then the dose could be titrated up. Initially, participants were allowed to titrate to doses up to 25 mg, however, the maximum dose was then limited to 10 mg.
- Overall LTSE OCA: After completion of the 12-month DB phase, all participants were offered the opportunity to enter an open-label LTSE for up to 5 years beginning at 5 mg OCA, and then the dose could be titrated up. Initially, participants were allowed to titrate to doses up to 25 mg, however, the maximum dose was then limited to 10 mg.
Arm/Group | DB 5-10 mg | DB OCA 10 mg | DB Placebo | LTSE OCA (DB OCA 5-10 mg) | LTSE OCA (DB 10 mg) | LTSE OCA (DB Placebo) | Overall LTSE OCA
Serious Adverse Events (participants affected / at risk) | 11/70 | 8/73 | 3/73 | 30/63 | 19/64 | 20/66 | 69/193
Other Adverse Events (participants affected / at risk) | 64/70 | 64/73 | 62/73 | 61/63 | 62/64 | 64/66 | 187/193
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | DB 5-10 mg (N=70) | DB OCA 10 mg (N=73) | DB Placebo (N=73) | LTSE OCA (DB OCA 5-10 mg) (N=63) | LTSE OCA (DB 10 mg) (N=64) | LTSE OCA (DB Placebo) (N=66) | Overall LTSE OCA (N=193)
Anaemia (Blood and lymphatic system disorders) | 0 (0) | 1 (1) | 0 (0) | 2 (4) | 0 (0) | 0 (0) | 2 (4)
Splenic infarction (Blood and lymphatic system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (1)
Aortic valve stenosis (Cardiac disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1)
Atrial fibrillation (Cardiac disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 0 (0) | 2 (2)
Cardiac failure (Cardiac disorders) | 1 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1)
Cardiac failure congestive (Cardiac disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1)
Cardiomyopathy (Cardiac disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 1 (1)
Myocardial infarction (Cardiac disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (1)
Sick sinus syndrome (Cardiac disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Ventricular fibrillation (Cardiac disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1)
Cataract (Eye disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1)
Abdominal distension (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1)
Abdominal pain (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (1)
Abdominal pain lower (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 1 (1)
Abdominal wall haematoma (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 2 (2)
Ascites (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1)
Constipation (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1)
Haematemesis (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 1 (1)
Lower gastrointestinal haemorrhage (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1)
Oedematous pancreatitis (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1)
Oesophageal varices haemorrhage (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 1 (1) | 1 (1) | 4 (4)
Pancreatitis (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 2 (2)
Rectal prolapse (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 1 (1)
Splenic artery aneurysm (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0) | 1 (3) | 0 (0) | 0 (0) | 1 (3)
Upper gastrointestinal haemorrhage (Gastrointestinal disorders) | 1 (1) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 1 (1)
Varices oesophageal (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (2) | 1 (1) | 0 (0) | 0 (0) | 1 (1)
Volvulus (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 1 (1)
Chest pain (General disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Non-cardiac chest pain (General disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Oedema (General disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Polyserositis (General disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1)
Cholecystitis acute (Hepatobiliary disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (1)
Cholelithiasis (Hepatobiliary disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 1 (1)
Hepatic failure (Hepatobiliary disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 1 (1)
Hyperplastic cholecystopathy (Hepatobiliary disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 1 (1)
Jaundice (Hepatobiliary disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 1 (1)
Appendicitis (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 1 (1)
Bacterial sepsis (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1)
Cellulitis (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 1 (1)
Endocarditis (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (1)
Erysipelas (Infections and infestations) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Parotitis (Infections and infestations) | 1 (1) | 0 (0) | 0 (0) | 1 (3) | 0 (0) | 0 (0) | 1 (3)
Pneumonia (Infections and infestations) | 0 (0) | 1 (1) | 0 (0) | 3 (3) | 1 (1) | 0 (0) | 4 (4)
Postoperative wound infection (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (1)
Pyelonephritis (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1)
Pyelonephritis chronic (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (1)
Sepsis (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (1)
Urosepsis (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 1 (1)
Vaginal infection (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 1 (1)
Anastomotic ulcer (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 1 (1)
Ankle fracture (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 1 (1)
Clavicle fracture (Injury, poisoning and procedural complications) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (1)
Foot fracture (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1)
Ligament rupture (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 1 (1)
Lower limb fracture (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 1 (1)
Meniscus lesion (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 1 (1)
Post procedural haemorrhage (Injury, poisoning and procedural complications) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 2 (2)
Procedural pain (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 2 (2)
Radius fracture (Injury, poisoning and procedural complications) | 0 (0) | 1 (2) | 0 (0) | 2 (2) | 2 (3) | 0 (0) | 4 (5)
Rib fracture (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 1 (2) | 0 (0) | 0 (0) | 1 (2)
Spinal compression fracture (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1)
Tibia fracture (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 1 (1)
Wrist fracture (Injury, poisoning and procedural complications) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (1)
Medical observation (Investigations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1)
Hypoglycaemia (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1)
Hyponatraemia (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 1 (1)
Haemarthrosis (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 1 (1)
Intervertebral disc protrusion (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (1)
Osteoarthritis (Musculoskeletal and connective tissue disorders) | 0 (0) | 2 (2) | 0 (0) | 2 (2) | 5 (6) | 0 (0) | 7 (8)
Rotator cuff syndrome (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 1 (1)
Spondylolisthesis (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1)
Systemic sclerosis (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 1 (1)
Basal cell carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1)
Breast cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1)
Chronic myeloid leukaemia (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1)
Chronic obstructive pulmonary disease (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1)
Colorectal cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 1 (1)
Hepatic neoplasm malignant (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1)
Hepatic neoplasm malignant recurrent (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1)
Lip neoplasm malignant stage unspecified (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1)
Renal oncocytoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1)
Uterine leiomyoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 1 (1)
Carpal tunnel syndrome (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1)
Hepatic encephalopathy (Nervous system disorders) | 1 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Ischaemic stroke (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 1 (1)
Loss of consciousness (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1)
Syncope (Nervous system disorders) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 2 (2)
Transient ischaemic attack (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 1 (1)
Depression (Psychiatric disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (1)
Major depression (Psychiatric disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (1)
Nephrolithiasis (Renal and urinary disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (1)
Nephropathy toxic (Renal and urinary disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1)
Renal atrophy (Renal and urinary disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 1 (1)
Renal failure (Renal and urinary disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1)
Renal failure acute (Renal and urinary disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (1)
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Interstitial lung disease (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Neurodermatitis (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (1)
Hypertension (Vascular disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 1 (1)
Intra-abdominal haematoma (Vascular disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (1)
Temporal arteritis (Vascular disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (1)
Varicose vein (Vascular disorders) | 2 (2) | 0 (0) | 0 (0) | 2 (2) | 0 (0) | 0 (0) | 2 (2)
OTHER ADVERSE EVENTS (reported when occurring in more than 4.50% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | DB 5-10 mg (N=70) | DB OCA 10 mg (N=73) | DB Placebo (N=73) | LTSE OCA (DB OCA 5-10 mg) (N=63) | LTSE OCA (DB 10 mg) (N=64) | LTSE OCA (DB Placebo) (N=66) | Overall LTSE OCA (N=193)
Pruritus (Skin and subcutaneous tissue disorders) | 39 (93) | 50 (99) | 28 (49) | 49 (249) | 51 (198) | 50 (180) | 150 (627)
Rash (Skin and subcutaneous tissue disorders) | 3 (3) | 4 (4) | 3 (3) | 7 (9) | 5 (5) | 2 (2) | 14 (16)
Eczema (Skin and subcutaneous tissue disorders) | 4 (4) | 2 (2) | 0 (0) | 5 (5) | 4 (4) | 5 (7) | 14 (16)
Nasopharyngitis (Infections and infestations) | 17 (27) | 13 (15) | 13 (19) | 23 (66) | 23 (39) | 11 (22) | 57 (127)
Urinary tract infection (Infections and infestations) | 4 (6) | 4 (6) | 8 (15) | 17 (31) | 19 (27) | 15 (23) | 51 (81)
Upper respiratory tract infection (Infections and infestations) | 4 (4) | 4 (4) | 8 (8) | 12 (21) | 11 (17) | 11 (16) | 34 (54)
Influenza (Infections and infestations) | 5 (5) | 4 (4) | 4 (5) | 12 (17) | 12 (17) | 10 (17) | 34 (51)
Sinusitis (Infections and infestations) | 1 (1) | 4 (5) | 0 (0) | 7 (7) | 9 (11) | 8 (11) | 24 (29)
Bronchitis (Infections and infestations) | 4 (4) | 1 (1) | 0 (0) | 7 (7) | 7 (7) | 6 (10) | 20 (24)
Nausea (Gastrointestinal disorders) | 4 (5) | 8 (10) | 9 (18) | 14 (20) | 13 (19) | 10 (15) | 37 (54)
Diarrhoea (Gastrointestinal disorders) | 2 (3) | 8 (10) | 8 (13) | 8 (15) | 11 (17) | 14 (26) | 33 (58)
Abdominal pain upper (Gastrointestinal disorders) | 5 (5) | 4 (5) | 5 (8) | 9 (12) | 10 (11) | 12 (13) | 31 (36)
Constipation (Gastrointestinal disorders) | 5 (5) | 5 (5) | 4 (7) | 12 (12) | 9 (9) | 7 (8) | 28 (29)
Abdominal distension (Gastrointestinal disorders) | 3 (3) | 3 (3) | 7 (7) | 5 (7) | 7 (7) | 5 (5) | 17 (19)
Dyspepsia (Gastrointestinal disorders) | 4 (4) | 0 (0) | 8 (11) | 7 (12) | 8 (8) | 5 (5) | 20 (25)
Vomiting (Gastrointestinal disorders) | 3 (3) | 3 (3) | 5 (8) | 5 (7) | 7 (9) | 2 (2) | 14 (18)
Gastrooesophageal reflux disease (Gastrointestinal disorders) | 2 (2) | 4 (5) | 4 (6) | 7 (7) | 9 (12) | 4 (4) | 20 (23)
Abdominal pain (Gastrointestinal disorders) | 3 (3) | 1 (1) | 6 (6) | 11 (15) | 7 (9) | 8 (8) | 26 (32)
Abdominal discomfort (Gastrointestinal disorders) | 5 (5) | 0 (0) | 1 (5) | 5 (5) | 0 (0) | 2 (2) | 7 (7)
Fatigue (General disorders) | 11 (13) | 17 (25) | 10 (12) | 24 (46) | 24 (43) | 15 (20) | 63 (109)
Oedema peripheral (General disorders) | 2 (2) | 5 (7) | 2 (3) | 10 (15) | 8 (12) | 8 (10) | 26 (37)
Pyrexia (General disorders) | 0 (0) | 5 (6) | 1 (1) | 5 (6) | 6 (8) | 5 (5) | 16 (19)
Back pain (Musculoskeletal and connective tissue disorders) | 4 (4) | 4 (5) | 8 (8) | 10 (13) | 11 (15) | 10 (10) | 31 (38)
Arthralgia (Musculoskeletal and connective tissue disorders) | 4 (5) | 7 (7) | 3 (3) | 14 (17) | 17 (23) | 15 (18) | 46 (58)
Muscle spasms (Musculoskeletal and connective tissue disorders) | 2 (2) | 2 (2) | 4 (5) | 4 (4) | 4 (7) | 3 (3) | 11 (14)
Headache (Nervous system disorders) | 12 (26) | 6 (7) | 13 (16) | 20 (43) | 15 (22) | 9 (10) | 44 (75)
Cough (Respiratory, thoracic and mediastinal disorders) | 4 (5) | 6 (6) | 5 (9) | 12 (23) | 11 (16) | 12 (16) | 35 (55)
Oropharyngeal pain (Respiratory, thoracic and mediastinal disorders) | 5 (5) | 6 (8) | 1 (1) | 6 (6) | 8 (11) | 4 (6) | 18 (23)
Insomnia (Psychiatric disorders) | 2 (2) | 3 (3) | 7 (8) | 6 (6) | 7 (7) | 7 (11) | 20 (24)
Dry eye (Eye disorders) | 2 (3) | 4 (4) | 4 (4) | 3 (4) | 10 (11) | 2 (2) | 15 (17)
Anaemia (Blood and lymphatic system disorders) | 2 (2) | 3 (3) | 4 (5) | 8 (12) | 7 (8) | 4 (5) | 19 (25)
Palpitations (Cardiac disorders) | 2 (3) | 5 (5) | 1 (1) | 4 (6) | 5 (5) | 2 (2) | 11 (13)
Procedural pain (Injury, poisoning and procedural complications) | 4 (4) | 1 (1) | 1 (3) | 8 (9) | 4 (5) | 4 (7) | 16 (21)
Hypothyroidism (Endocrine disorders) | 4 (4) | 1 (1) | 1 (1) | 4 (4) | 3 (3) | 3 (3) | 10 (10)
Osteopenia (Musculoskeletal and connective tissue disorders) | 1 (1) | 1 (1) | 0 (0) | 9 (9) | 6 (6) | 6 (7) | 21 (22)
Pain in extremity (Musculoskeletal and connective tissue disorders) | 3 (3) | 1 (1) | 3 (3) | 7 (11) | 5 (5) | 8 (9) | 20 (25)
Hypertension (Vascular disorders) | 0 (0) | 2 (2) | 1 (1) | 5 (6) | 6 (7) | 8 (8) | 19 (21)
Osteoarthritis (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1) | 1 (1) | 4 (5) | 6 (8) | 5 (7) | 15 (20)
Dizziness (Nervous system disorders) | 3 (5) | 2 (2) | 2 (2) | 5 (9) | 7 (7) | 2 (2) | 14 (18)
Skin lesion (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1) | 3 (3) | 3 (5) | 5 (7) | 6 (8) | 14 (20)
Depression (Psychiatric disorders) | 1 (1) | 1 (1) | 0 (0) | 5 (6) | 5 (6) | 3 (4) | 13 (16)
Myalgia (Musculoskeletal and connective tissue disorders) | 1 (1) | 3 (3) | 0 (0) | 4 (5) | 7 (9) | 2 (2) | 13 (16)
Respiratory tract infection (Infections and infestations) | 0 (0) | 0 (0) | 3 (3) | 5 (6) | 4 (5) | 4 (5) | 13 (16)
Cystitis (Infections and infestations) | 1 (2) | 2 (2) | 0 (0) | 5 (12) | 5 (15) | 2 (3) | 12 (30)
Herpes zoster (Infections and infestations) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 7 (8) | 4 (4) | 12 (13)
Musculoskeletal pain (Musculoskeletal and connective tissue disorders) | 1 (1) | 1 (1) | 1 (1) | 4 (5) | 5 (6) | 3 (3) | 12 (14)
Neck pain (Musculoskeletal and connective tissue disorders) | 1 (1) | 2 (2) | 1 (2) | 3 (3) | 4 (4) | 5 (5) | 12 (12)
Pneumonia (Infections and infestations) | 0 (0) | 2 (2) | 0 (0) | 2 (2) | 5 (8) | 5 (6) | 12 (16)
Asthenia (General disorders) | 2 (2) | 1 (1) | 1 (1) | 2 (2) | 3 (7) | 6 (6) | 11 (15)
Dry mouth (Gastrointestinal disorders) | 2 (2) | 3 (3) | 2 (2) | 3 (4) | 5 (5) | 3 (3) | 11 (12)
Gastritis (Gastrointestinal disorders) | 1 (1) | 1 (1) | 0 (0) | 2 (2) | 6 (7) | 3 (3) | 11 (12)
Haemorrhoids (Gastrointestinal disorders) | 0 (0) | 0 (0) | 2 (2) | 5 (6) | 1 (1) | 5 (5) | 11 (12)
Influenza like illness (General disorders) | 1 (1) | 3 (4) | 1 (1) | 4 (4) | 6 (9) | 1 (1) | 11 (14)
Osteoporosis (Musculoskeletal and connective tissue disorders) | 1 (1) | 1 (1) | 2 (2) | 2 (2) | 4 (5) | 5 (6) | 11 (13)
Varices oesophageal (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0) | 8 (8) | 2 (3) | 1 (1) | 11 (12)
Ascites (Gastrointestinal disorders) | 1 (1) | 1 (1) | 0 (0) | 6 (9) | 1 (1) | 3 (4) | 10 (14)
Cholelithiasis (Hepatobiliary disorders) | 2 (2) | 0 (0) | 0 (0) | 5 (6) | 4 (4) | 1 (1) | 10 (11)
Contusion (Injury, poisoning and procedural complications) | 3 (3) | 2 (3) | 2 (2) | 2 (2) | 5 (5) | 3 (3) | 10 (10)
Gastroenteritis (Infections and infestations) | 3 (3) | 1 (1) | 0 (0) | 4 (4) | 1 (1) | 5 (6) | 10 (11)
Toothache (Gastrointestinal disorders) | 0 (0) | 1 (1) | 1 (1) | 2 (2) | 5 (6) | 3 (3) | 10 (11)
Dental caries (Gastrointestinal disorders) | 2 (2) | 0 (0) | 0 (0) | 4 (5) | 1 (1) | 4 (6) | 9 (12)
Dry skin (Skin and subcutaneous tissue disorders) | 1 (1) | 2 (2) | 1 (1) | 1 (1) | 3 (3) | 5 (5) | 9 (9)
Sciatica (Nervous system disorders) | 0 (0) | 1 (1) | 0 (0) | 3 (3) | 3 (4) | 3 (4) | 9 (11)
Bone pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 3 (3) | 1 (1) | 5 (5)
Depressed mood (Psychiatric disorders) | 0 (0) | 1 (2) | 0 (0) | 0 (0) | 4 (5) | 1 (2) | 5 (7)
Dermatitis (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0) | 0 (0) | 3 (5) | 0 (0) | 2 (7) | 5 (12)
Diverticulum (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 3 (3) | 0 (0) | 5 (5)
Ear infection (Infections and infestations) | 0 (0) | 1 (1) | 1 (1) | 1 (1) | 1 (2) | 3 (3) | 5 (6)
Hepatic enzyme increased (Investigations) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 3 (5) | 1 (1) | 5 (7)
Hiatus hernia (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 3 (3) | 1 (1) | 5 (5)
Iron deficiency anaemia (Blood and lymphatic system disorders) | 0 (0) | 1 (1) | 0 (0) | 1 (4) | 1 (1) | 3 (4) | 5 (9)
Nasal congestion (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 2 (2) | 0 (0) | 3 (3) | 2 (2) | 0 (0) | 5 (5)
Oral herpes (Infections and infestations) | 1 (1) | 1 (1) | 1 (1) | 3 (4) | 1 (1) | 1 (1) | 5 (6)
Portal hypertensive gastropathy (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 3 (3) | 0 (0) | 2 (2) | 5 (5)
Rib fracture (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 3 (3) | 2 (2) | 0 (0) | 5 (5)
Thrombocytopenia (Blood and lymphatic system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 3 (3) | 2 (2) | 5 (5)
Urticaria (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 2 (3) | 1 (1) | 3 (4) | 1 (4) | 5 (9)
Arthropod bite (Injury, poisoning and procedural complications) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 4 (4) | 4 (4)
Bradycardia (Cardiac disorders) | 0 (0) | 0 (0) | 0 (0) | 3 (3) | 0 (0) | 1 (1) | 4 (4)
Excoriation (Injury, poisoning and procedural complications) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 3 (3) | 0 (0) | 4 (4)
Gastric polyps (Gastrointestinal disorders) | 0 (0) | 2 (2) | 0 (0) | 1 (1) | 3 (4) | 0 (0) | 4 (5)
Hepatomegaly (Hepatobiliary disorders) | 0 (0) | 0 (0) | 0 (0) | 3 (3) | 0 (0) | 1 (1) | 4 (4)
Low density lipoprotein increased (Investigations) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 3 (4) | 4 (5)
Night sweats (Skin and subcutaneous tissue disorders) | 3 (3) | 0 (0) | 0 (0) | 3 (3) | 0 (0) | 1 (1) | 4 (4)
Plantar fasciitis (Musculoskeletal and connective tissue disorders) | 0 (0) | 2 (2) | 0 (0) | 0 (0) | 3 (4) | 1 (1) | 4 (5)
Rash pruritic (Skin and subcutaneous tissue disorders) | 0 (0) | 2 (2) | 0 (0) | 0 (0) | 3 (3) | 1 (1) | 4 (4)
Gamma-glutamyltransferase increased (Investigations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 3 (3) | 3 (3)
Hyperhidrosis (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0) | 2 (2) | 3 (3) | 0 (0) | 0 (0) | 3 (3)
Hypoaesthesia (Nervous system disorders) | 1 (1) | 0 (0) | 0 (0) | 3 (5) | 0 (0) | 0 (0) | 3 (5)
Ligament rupture (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 3 (3) | 3 (3)
Tendon rupture (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 3 (3) | 0 (0) | 3 (3)
Scratch (Injury, poisoning and procedural complications) | 1 (1) | 3 (4) | 0 (0) | 1 (1) | 6 (7) | 2 (3) | 9 (11)
Conjunctivitis (Eye disorders) | 1 (1) | 2 (2) | 2 (2) | 2 (4) | 5 (6) | 1 (1) | 8 (11)
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 2 (3) | 0 (0) | 3 (4) | 3 (4) | 2 (3) | 3 (5) | 8 (12)
Erythema (Skin and subcutaneous tissue disorders) | 1 (1) | 3 (3) | 0 (0) | 2 (4) | 3 (4) | 3 (4) | 8 (12)
Fall (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 4 (4) | 0 (0) | 4 (4) | 8 (8)
Hypercholesterolaemia (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 2 (2) | 3 (4) | 2 (2) | 3 (3) | 8 (9)
Hypotension (Vascular disorders) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 2 (3) | 4 (4) | 8 (9)
Joint swelling (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 3 (3) | 1 (1) | 4 (4) | 8 (8)
Vertigo (Ear and labyrinth disorders) | 1 (1) | 0 (0) | 0 (0) | 4 (7) | 2 (2) | 2 (2) | 8 (11)
Vitamin D deficiency (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 1 (1) | 2 (2) | 3 (3) | 3 (3) | 8 (8)
Anxiety (Psychiatric disorders) | 2 (3) | 0 (0) | 2 (3) | 3 (5) | 1 (1) | 3 (3) | 7 (9)
Cardiac murmur (Cardiac disorders) | 0 (0) | 1 (1) | 0 (0) | 3 (3) | 2 (2) | 2 (2) | 7 (7)
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 1 (1) | 3 (3) | 1 (1) | 4 (6) | 2 (2) | 7 (9)
Hepatic cirrhosis (Hepatobiliary disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 2 (2) | 4 (4) | 7 (7)
Meniscus lesion (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 1 (2) | 5 (5) | 1 (1) | 7 (8)
Paraesthesia (Nervous system disorders) | 1 (1) | 1 (1) | 1 (1) | 2 (3) | 2 (2) | 3 (3) | 7 (8)
Rectal haemorrhage (Gastrointestinal disorders) | 0 (0) | 2 (2) | 0 (0) | 1 (1) | 2 (2) | 4 (4) | 7 (7)
Seasonal allergy (Immune system disorders) | 2 (2) | 1 (1) | 2 (2) | 4 (4) | 2 (2) | 1 (1) | 7 (7)
Splenomegaly (Blood and lymphatic system disorders) | 0 (0) | 0 (0) | 0 (0) | 4 (5) | 2 (2) | 1 (1) | 7 (8)
Tooth infection (Infections and infestations) | 1 (2) | 0 (0) | 0 (0) | 2 (3) | 3 (3) | 2 (2) | 7 (8)
Atrial fibrillation (Cardiac disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 3 (7) | 2 (2) | 6 (10)
Cataract (Eye disorders) | 0 (0) | 1 (1) | 0 (0) | 2 (2) | 3 (4) | 1 (1) | 6 (7)
Diabetes mellitus (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 3 (3) | 3 (5) | 6 (8)
Ear pain (Ear and labyrinth disorders) | 2 (2) | 0 (0) | 1 (1) | 2 (3) | 3 (3) | 1 (1) | 6 (7)
Lower respiratory tract infection (Infections and infestations) | 2 (2) | 0 (0) | 1 (1) | 4 (8) | 1 (2) | 1 (5) | 6 (15)
Pharyngitis (Infections and infestations) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 3 (6) | 2 (2) | 6 (9)
Renal cyst (Renal and urinary disorders) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 3 (3) | 1 (1) | 6 (6)
Sleep disorder (Psychiatric disorders) | 3 (7) | 0 (0) | 0 (0) | 3 (8) | 1 (1) | 2 (2) | 6 (11)
Weight decreased (Investigations) | 0 (0) | 0 (0) | 0 (0) | 3 (3) | 2 (2) | 1 (1) | 6 (6)
Abdominal pain lower (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0) | 3 (4) | 1 (1) | 1 (1) | 5 (6)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Principal Investigators must wait 18 months after the study ends to publish their results and a multi-center publication must come first. The sponsor has a 45 day review period with the option to extend to an additional 90 days.